CLINICAL TRIAL: NCT03127579
Title: Family Meal Duration and Children's Eating Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max Planck Institute for Human Development (Other)
Collaborators: University of Mannheim (Other)
Responsible Party: Principal Investigator, Mattea Dallacker, Principle Investigator, Max Planck Institute for Human Development
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ARC1
Record Dates: First submitted 2016-11-17; First posted 2017-04-25 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Feeding Behavior; Eating; Child Behavior; Family Relations
MeSH Terms: conditions — Feeding Behavior; Child Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Longer meal duration (Experimental): Families eat longer as they usually do
  Interventions: Behavioral: Longer meal duration
- Usual meal duration (No Intervention): Families eat as long as they usually do

INTERVENTIONS:
Behavioral: Longer meal duration — Participants have 50% more time to eat than usual
  Arms: Longer meal duration

SUMMARY:
The goal of this study is to test whether a longer meal duration could improve the diet quality of children. To answer this question we want to take an experimental approach by implementing a longer family meal duration to examine differences in children's eating behavior. The family dinner within a laboratory setting will be video taped and the main outcome is children's fruit and vegetables consumption.

DETAILED DESCRIPTION:
Parent-child pairs have two dinner in a laboratory setting. The study design is a within-subject design: In the control condition they have as much time as they usual. In the intervention condition they have 50% more time than usual. Order of the two condition is counter balanced. The lab dinner reflects a typical German dinner which consists of bread, cheese, cold meat and fruits and vegetables. Additionally a dessert is served after the main meal. The foods served reflect food preferences of the child. All dinners are video taped. Key outcome variables are consumption of fruits and vegetables, dessert, eating rate and amount time engaged in positive and negative social interaction

ELIGIBILITY:
Inclusion Criteria:

* children and their nutritional gatekeeper

Exclusion Criteria:

* food allergies
* participants follow special diet

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Food consumption | Food intake is measured during the lab meal
  The lab dinner is video taped. Consumption of fruits, vegetables, bread, cheese, cold meat and dessert (cookies or pudding), drinks (water, or milk, or juice) are coded by two independent rater.

SECONDARY OUTCOMES:
Social interactions: positive and negative communication | Social interaction is measured during the lab meal
  The lab dinner is video taped. Social interactions are coded according to the ABC family mealtime coding system by Fiese, Winter & Botti, 2011.
Eating rate | From the start to the end of the meal (about 20-30 minutes)
  Bites per minute coded from video tapes
Hunger | Participants filled out a questionnaire 5 minutes after the lab dinner
  Hunger rating scale (ranging from 1= I am really hungry to 5 = I am not hungry at all)
Atmosphere | Participants filled out a questionnaire 5 minutes after the lab dinner
  Atmosphere rating scale (ranging from 1= very negative to 5 = very positive)

CONTACTS AND LOCATIONS:
Locations (1):
- Max Planck Institute for Human Development, Berlin, Germany

REFERENCES:
- [Derived] Dallacker M, Knobl V, Hertwig R, Mata J. Effect of Longer Family Meals on Children's Fruit and Vegetable Intake: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e236331. doi: 10.1001/jamanetworkopen.2023.6331. PMID 37010871